CLINICAL TRIAL: NCT06964178
Title: The Effect of Antimicrobial Photodynamic Therapy on the Healing of the Post-extraction Socket of the Mandibular Third Molar: a Randomized Clinical Study
Brief Title: The Effect of Photodynamic Therapy on Post-extraction Third Molar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Alessia Pardo, PhD, Dental Hygienist, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Univr4242
Record Dates: First submitted 2025-04-23; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Photodynamic Therapy; Third Molar Extraction; Antimicrobial Photodynamic Therapy
Keywords: Photodynamic Therapy; third molar extraction; Soft tissue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- antimicrobial photodynamic therapy (aPDT) after extraction of third molar (Experimental): extraction, the need for osteotomy, odontotomy, and root separation was recorded. The test group received antimicrobial photodynamic therapy (aPDT) immediately before suturing. A diode laser with a wavelength of 660 nm was used (Helbo® TheraLite Laser, Bredent, Germany). a wavelength of 660 nm was used (Helbo® TheraLite Laser, Bredent, Germany). A strip of gauze was soaked with Helbo® Biofilm Marker and the socket was swabbed. This liquid is based on phenothiazine chloride and was provided in pre-packaged sterile syringes. Photosensitizer was left in the post-extraction socket for three minutes. All alveolar walls were irradiated for ten seconds each (disto-lingual, lingual, mesio-lingual, mesio-buccal, buccal, disto-buccal), for a total duration of 60 seconds.
  Interventions: Device: Experimental: antimicrobial photodynamic therapy (aPDT) after extraction of third molar
- extraction of third molar (No Intervention): A trapezoidal flap was elevated, and the tooth was extracted. During the extraction, the need for the post-extraction socket was sutured with Vicryl 4.0 sutures. In the control group, once the tooth was removed, the post-extraction site was cleaned by curettage, washed with saline, and then sutured with Vicryl 4.0 suture. The duration of the surgery was recorded, as well as the degree of intraoperative bleeding., odontotomy, and root separation was recorded.

INTERVENTIONS:
Device: Experimental: antimicrobial photodynamic therapy (aPDT) after extraction of third molar — In the test, a photoactive substance activated with laser light (20 mW, 660 nm) was applied to the post-extraction site for 60 seconds before suturing, to promote healing and disinfection
  Other Names: antimicrobial photodynamic therapy (aPDT) after extraction of third molar
  Arms: antimicrobial photodynamic therapy (aPDT) after extraction of third molar

SUMMARY:
The extraction of lower third molars is one of the most frequent procedures in oral surgery. For this reason, the extraction of these teeth generally requires a surgical approach involving the elevation of a mucoperiosteal flap and osteotomy to allow the use of elevators and removal of tooth in pieces or as a whole depending on the situation. As a result, it is a more invasive procedure than simple dental extraction, which leads a more challenging healing period for the patient, with complications such as pain, swelling, and trismus. Literature studies suggest that the peak of pain reported by patients occurs 3-5 hours after the local anesthetic wears off, while swelling reaches its maximum in the first 24-48 hours before gradually decreasing. In the first hours following the surgery, in addition to symptom onset, reparative mechanisms begin, contributing to the healing of the post-extraction site. Independent of the use of bone grafts, antimicrobial photodynamic therapy (aPDT) has been introduced to enhance healing and for disinfection of the extraction site5,6. aPDT uses a non-thermal photochemical reaction which promotes the excitation of a nontoxic dye (photosensitizer) by light at an appropriate wavelength. This causes an interaction with molecular oxygen and acts by damaging biomolecules selectively and destroying bacterial membranes7. The efficacy of this therapy in reducing bacterial load has been demonstrated in literature, and it has been widely used in patients with periodontitis or peri-implantitis since several years8. Although the primary use of antimicrobial photodynamic therapy seems to be related to periodontal and peri-implant diseases, its use in oral surgery to disinfect the socket and reduce the risk of complications related to bacterial contamination of the surgical site should not be underestimated9. Furthermore, the biostimulator effect of the laser can promote tissue healing after surgery through vasodilation, activation of microcirculation, and enhancement of tissue metabolism, thus reducing the recovery time for the patient10. There are still a few papers in literature that evaluate the effect of aPDT on post-operative healing after wisdom tooth extractions. This study aimed to investigate the effect of aPDT on the healing of soft and hard tissues and on post-surgical discomfort in subjects undergoing mandibular third molar extraction. The null hypothesis is that aPDT has no beneficial effects compared to spontaneous healing.

DETAILED DESCRIPTION:
Patients in need of unilateral mandibular third molar extraction were randomly assigned to test or control group before surgery. In the test, a photoactive substance activated with laser light (20 mW, 660 nm) was applied to the post-extraction site for 60 seconds before suturing, to promote healing and disinfection. The control group did not receive any laser applications after tooth removal.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients (ASA I/II according to the American Society of Anesthesiologists classification),
* Requiring at least one mandibular third molar extraction without preoperative significant pain or edema
* Patients aged between 14-39 years.

Exclusion Criteria:

* Patients with systemic diseases interfering with normal healing process
* Pregnant or lactating women
* Patients with third molar buds
* Patients with continuity between the roots of the lower third molar
* The cortical bone of the mandibular nerve canal were excluded from the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-11-03 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Probing Pocket Depth PPD Index | T0 (Baseline), T1(14 days after extraction) and T2 (3 month after extraction)
  Probing depth is the distance from the gingival margin to the base of the pocket (mm)

SECONDARY OUTCOMES:
Recession REC Index | T0 (Baseline), T1(14 days after extraction) and T2 (3 month after extraction)
  Recession is the apical shift of the marginal tissues associated with the attachment loss exposing the root or implant surface to the oral environment (mm)
Clinical attachment level CAL Index | T0 (Baseline), T1(14 days after extraction) and T2 (3 month after extraction)
  measured in mm as distance from the CEJ to the gingival margin (GM)
Plaque Index | T0 (Baseline), T1(14 days after extraction) and T2 (3 month after extraction)
  This index ascertains the thickness of plaque along the gingival margin (%)
Bleeding on probing BOP Index | T0 (Baseline), T1(14 days after extraction) and T2 (3 month after extraction)
  is an indicator of tissue inflammatory response to bacterial pathogens (%)
Landry's healing index | T0 (Baseline), T1(14 days after extraction) and T2 (3 month after extraction)
  (code 1 (very poor healing); • code 2 (poor healing); • code 3 (good healing) ; • code 4 (very good healing); • code 5 (excellent healing)
Bone density Index | T0 (Baseline), T1(14 days after extraction) and T2 (3 month after extraction)
  bone density through intraoral radiographs was also assessed through peri-apical x-rays at T2, attributing a value from 0 to 2. A value of 0 corresponded to a low degree of bone density, with radiolucency in correspondence with the extracted dental element and marked radiopacity; a value of 1 corresponded to a medium density with slight radiopacity at the extracted third molar, compatible with the apposition of new immature bone and persistence of marked radiopacity; a value of 2 corresponded to a high bone density with radiopacity in correspondence with the extracted element, compatible with new bone apposition..

CONTACTS AND LOCATIONS:
Locations (1):
- Alessia Pardo, Verona, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomized trials. Ann Intern Med. 2010 Jun 1;152(11):726-32. doi: 10.7326/0003-4819-152-11-201006010-00232. Epub 2010 Mar 24. PMID 20335313
- [Background] Yamada SI, Hasegawa T, Yoshimura N, Hakoyama Y, Nitta T, Hirahara N, Miyamoto H, Yoshimura H, Ueda N, Yamamura Y, Okuyama H, Takizawa A, Nakanishi Y, Iwata E, Akita D, Itoh R, Kubo K, Kondo S, Hata H, Koyama Y, Miyamoto Y, Nakahara H, Akashi M, Kirita T, Shibuya Y, Umeda M, Kurita H. Prevalence of and risk factors for postoperative complications after lower third molar extraction: A multicenter prospective observational study in Japan. Medicine (Baltimore). 2022 Aug 12;101(32):e29989. doi: 10.1097/MD.0000000000029989. PMID 35960058
- [Background] Fraga RS, Antunes LAA, Fialho WLS, Valente MI, Gomes CC, Fontes KBFC, Antunes LS. Do Antimicrobial Photodynamic Therapy and Low-Level Laser Therapy Minimize Postoperative Pain and Edema After Molar Extraction? J Oral Maxillofac Surg. 2020 Dec;78(12):2155.e1-2155.e10. doi: 10.1016/j.joms.2020.08.002. Epub 2020 Aug 7. PMID 32890472
- [Background] Souza MRJ, Meyfarth S, Fraga RS, Fontes KBFC, Guimaraes LS, Antunes LAA, Antunes LS. Do Antimicrobial Photodynamic Therapy and Low-Level Laser Therapy Influence Oral Health-Related Quality of Life After Molar Extraction? J Oral Maxillofac Surg. 2023 Aug;81(8):1033-1041. doi: 10.1016/j.joms.2023.04.002. Epub 2023 Apr 13. PMID 37094757
- [Background] Schar D, Ramseier CA, Eick S, Arweiler NB, Sculean A, Salvi GE. Anti-infective therapy of peri-implantitis with adjunctive local drug delivery or photodynamic therapy: six-month outcomes of a prospective randomized clinical trial. Clin Oral Implants Res. 2013 Jan;24(1):104-10. doi: 10.1111/j.1600-0501.2012.02494.x. Epub 2012 May 9. PMID 22568744
- [Background] Fisher SE, Frame JW, Rout PG, McEntegart DJ. Factors affecting the onset and severity of pain following the surgical removal of unilateral impacted mandibular third molar teeth. Br Dent J. 1988 Jun 11;164(11):351-4. doi: 10.1038/sj.bdj.4806453. No abstract available. PMID 3165011